CLINICAL TRIAL: NCT03742128
Title: The REFUGE-study: Health and Quality of Life Among Resettled Syrian Refugees and Asylum-seekers in Norway (REFUGE-I)
Brief Title: Health and Quality of Life Among Resettled Syrians in Norway
Acronym: REFUGE-I
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Norwegian Center for Violence and Traumatic Stress Studies (Other)
Collaborators: Norwegian Institute of Public Health (Other Government); Inland Norway University of Applied Sciences (Other); Swedish Red Cross University College (Other); Karolinska Institutet (Other)
Responsible Party: Sponsor
Other Study IDs: NKVTS 2017/1252
Record Dates: First submitted 2018-11-12; First posted 2018-11-15 (Actual); Last update posted 2018-11-30 (Actual); Status verified 2018-11

CONDITIONS: Mental Health Impairment; Stress, Psychological; Quality of Life; Health, Subjective; Posttraumatic Stress Disorder; Anxiety; Depression
MeSH Terms: conditions — Stress, Psychological; Stress Disorders, Post-Traumatic; Anxiety Disorders; Depression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Brief summary The civil war in Syria has taken a severe toll on the Syrian population, with over 350 000 dead and more than 10 million Syrians forced to leave their home since 2011. The majority of the estimated 5.6 million Syrians who have left the country as refugees currently reside in Syria's neighboring countries (Turkey, Jordan and Lebanon), while about 1 million have fled to Europe. In the peak year of 2015, a little over 10500 Syrians applied for asylum in Norway and an estimated 26 000 lived in the country at the start of 2018 according to statistics from the Norwegian Directorate of Immigration.

Being a refugee or resettled refugee is psychologically stressful and increases the risk of ill mental health. Prior research has demonstrated high to very high levels of posttraumatic stress disorder (PTSD), depression and anxiety in refugees compared to normal populations. As highlighted in prior review articles on the subject, there is a lack of studies on refugees originating from the Middle Eastern countries, and there is a need for future studies on refugee mental health to move beyond the focus on PTSD, depression and anxiety in order to capture the wider psychological consequences associated with being a refugee or resettled refugee. With the current number of displaced people globally approaching an unprecedented 70 million, including more than 25 million refugees, the need to understand and address the health challenges in this population is more pressing than ever.

The present study, REFUGE-I, constitutes the first phase of a planned longitudinal cohort study (REFUGE-study) on health and quality of life among resettled Syrian refugees in Norway. The overarching aims of REFUGE-I are to recruit a representative sample of Syrian adults who are willing to participate in the longitudinal cohort study and to obtain baseline information on health-related topics as well as demographics for this recruited sample.

REFUGE-I will use a cross-sectional survey design. The study population will be a random and representative sample of 10 000 Syrians over 18 years who arrived in Norway between 2015 and 2017, and who currently live and have a registered residential address in Norway. The sampled group will be contacted and informed about the study through postal mail. Information about the study will also be distributed through other channels: regular media (e.g. television and newspapers), social media (e.g. Facebook), District Medical Doctors/Public Health Officers, and a study web-page with more detailed information on the study including instructive animation videos in Arabic. Those consenting to participate will be asked to fill out and return a postal survey questionnaire on demographics and health-related topics focusing on:

Symptoms of posttraumatic stress, anxiety and depression Quality of life Self-reported physical health (focusing on subjective pain) Sleep difficulties and alcohol consumption patterns Social support Potentially traumatic experiences before or during the flight from Syria Stress experienced after arrival in Norway (post-migratory stress)

Participants will also be asked whether the research group can contact them again for the second and third phase of the longitudinal study, and informed that consent to participation entails consent that survey data will be linked to Norwegian registry data on education, work participation and sick-leave, drug prescriptions and utilization of the health-care system. The registry data will be linked to survey data in the later phases of the larger longitudinal study.

The main objective of the REFUGE-I study is to obtain and publish a thorough cohort profile that includes descriptive statistics for the final sample on the above-listed health-related topics, as well as information and statistics on potential selection bias issues that might affect the generalizability of findings.

The study is a collaborative effort between five research institutions and universities in Norway and Sweden. One of the collaborating partners, The Swedish Red Cross University College, has already conducted a similar study on 1215 resettled adult Syrian refugees in Sweden, and results from REFUGE-I will be compared to the findings from the Swedish study. Moreover, an important long-term goal for the larger REFUGE-study is to help advance research on refugees by making resources from the study available online, and through the creation of a large database containing pooled data from the REFUGE-study and studies done through the Swedish Red Cross University College and potentially other national and international research groups.

DETAILED DESCRIPTION:
Participants:

A complete list of potential participants meeting Inclusion criteria (see relevant section in the submitted registration) was obtained in collaboration with the Norwegian National Registry administered by the Norwegian Tax Administration. The complete list consisted of 14350 individuals which constituted the study's sampling frame. A simple random probability sample of 10 000 individuals was selected from the sampling frame (sampling fraction = 0.7). The actual sampling was conducted without any involvement from members of the REFUGE-I research team.

Data collection:

All sampled participants will be sent a postal package to their registered residential address in Norway. The package will contain a prepaid return envelope, the survey questionnaire and a cover letter in Arabic describing the purpose of the study, its voluntary nature, what potential participants can expect if they do participate, and how issues surrounding confidentiality and anonymity will be handled. The cover letter also highlights that survey data will be linked to registry data as part of the longitudinal study. Potential participants will be enabled to give written informed consent to participation at the bottom of the cover letter and instructed to enclose the written consent with the completed survey questionnaire in the prepaid return envelope. Data from participants returning the questionnaire without also submitting written consent to participation will be deleted in accordance with agreements made with the Regional Committees for Medical and Health Research Ethics (REC) - Region South East which granted the ethical approval for the study.

The survey questionnaire is eight pages long and expected to take about an hour to complete. All instructions and questions in the questionnaire are in Arabic. Standard and pre-existing scales in Arabic were used whenever available and Arabic translations were done by professional translators in collaboration with an Arabic speaking reference group for scales/items that did not already exist in Arabic. Potential participants will have about 8 weeks to complete and return the questionnaire with written consent. One postal reminder, together with a blank copy of the survey questionnaire and a prepaid return envelope will be sent out to participants who have not returned the questionnaire by a preset deadline - about two weeks before the anticipated closing date for data collection (approximately January 15, 2019). This is in accordance with Norwegian rules and regulations governing research with voluntary subjects which prohibits more than one reminder being sent out.

Analysis:

Three main articles are stipulated to be submitted for publication from the data collected through the survey questionnaire of REFUGE-I. Article one will report descriptive statistics on the main outcome variables: depression; anxiety; and symptoms of posttraumatic stress disorder across key demographic and background variables in the sample, and describe the flow of participants and discuss potential selection bias issues. Article two will provide descriptive statistics on somatic pain, sleep difficulties and perceived general health, and report findings across the same demographic and background variables as article one and across the main outcomes of article one (depression, anxiety and symptoms of posttraumatic stress disorder). Article three will present statistics on reported quality of life across demographic and background variables, and across the outcome variables of article one and two.

Alternatively, one larger article will be submitted for publication incorporating all of the themes outlined in the three articles above.

Specific analysis plans for each article/theme are described below:

Article I:

Title: "Prevalence of common mental health disorders in adult Syrian refugees resettled in Norway between 2015 and 2017: a cross-sectional survey questionnaire study".

In order to compare results to a parallel study on newly resettled adult refugees in Sweden conducted by one of our collaborating institutions, Article I will use similar outcome and predictor variables as this study. The main outcome variables will be:

Prevalence of symptom-based posttraumatic stress disorder (PTSD) as measured through the first 16 items in the section on trauma symptoms (section IV) in the Harvard Trauma Questionnaire (HTQ). A mean-item score ≥ 2.06 will define a "checklist-positive" PTSD case. To be included in analyses, participants must have answered 14 or more of the 16 items on the HTQ scale.

Prevalence of symptom-based depression and anxiety as measured through the two subscales on depression and anxiety in the Hopkins Symptom Checklist (HSCL-25). A mean-item score ≥ 1.80 and ≥ 1.75 will define a "checklist-positive" depression and anxiety case, respectively. To be included in analyses, participants must have answered ≥ 23 items on the 25-item scale.

The outcome variables above will be summarized for the whole sample population and across the following demographic and background variables:

Gender Age; split into age groups: 18-29; 30-39; 40-49; 50-64; >64. Education; split into the categories: 0-9 years; 10-12 years; >12 years Civil status; split into the categories: Married; Unmarried; Divorced/separated/widow(er); Other Arrival status; split into the categories: Asylum seeker; Quota/resettlement refugee; Family immigration; Other Year of arrival/immigration to Norway; split into: 2015; 2016; 2017. Refugee trauma history measured through the Refugee Trauma History Checklist (RTHC). The two scales contained in this checklist will be combined - that is, the period will be "prior to arriving in Norway".

Post-migration stress measured through seven main items of the Post-migration stress scale thought to tap into the relevant domains of post-migration stress. Answers to each item will be dichotomized so that those answering "often" or "very often" are classified as having had this reaction often (i.e. positive for that post-migratory stress reaction)

Prevalence estimates will be presented with 95% confidence intervals (95% CIs). Odds ratios (ORs) with 95% CIs will be used when summarizing the main outcome variables across refugee trauma history and post-migration stress. More specifically, the odds of having a symptom-level above vs. below the preset cut-off value for the main outcomes will be calculated for each binary (Y/N) item on the trauma history and post-migration stress scales (eight and seven items for the two scales, respectively). The positive answer ("Yes") will define exposed for each item when reporting the ORs.

In addition, descriptive statistics on the prevalence of refugee-related possible traumatic events will be presented. Descriptive statistics (distribution, mean and variance) on the seven domains of the complete 24-item post-migration scale will be presented and compared to the study in Sweden. The prevalence of comorbidity between checklist-positive anxiety, depression and PTSD will also be reported with 95% CIs.

The number of participants contributing data to a specific statistics will be reported. The study will report, compare and discuss statistics on the participants vs. the sample frame on all available parameters for both groups in order to evaluate selection bias issues (anticipated available parameters include: age, gender, civil/marital status, permanent vs temporary residence status, number of registered mobile phone numbers).

Article II:

Title: "Subjective health and pain, and sleep difficulties in adult Syrian refugees resettled in Norway between 2015 and 2017: a cross-sectional survey questionnaire study".

Main outcomes:

Somatic pain (including pain in muscles and joints and general pain), measured as described under Outcome Measures. Statistics on pain in muscles and joints will be aggregated (i.e. all items will be combined) and reported as the percentage of participants in each of three categories: Not troubled with pain in muscles and joints (Not troubled reported for all items); Somewhat troubled with pain in muscles and joints (Somewhat troubled reported for at least one item); Very troubled with pain in muscles and joints (Very troubled for at least one item). Participants must have answered at least four of the five items (if all answers are Not troubled), or Somewhat troubled/Very troubled on at least one item to be included in analyses. Statistics on general pain will be presented in an identical manner (i.e. the percentage in each of three categories, aggregated across all items on general pain) Sleep difficulties, measured as described under Outcome Measures. The overall mean-item score will be reported, as well as the estimated prevalence of insomnia, defined by the following criteria: a score of 3 or above on at least one of the first 4 items + a score of 3 or higher on at least one of the last 2 items. Participants must have answered at least five of the six items to be included in analyses when analyzing the mean-item score of the scale. When analyzing the prevalence of insomnia, participants must have answered at least three of the first four items and one of the last two items; or, they must have a score of 3 or above on at least one of the first four items and a score of 3 or above on at least one of the last two items to be included in analyses.

Perceived general health, measured as described under Outcome Measures. Statistics on perceived general health will be reported as the percentage of participants in each answer category (with 95% CIs). Question one on overall health will be dichotomized with Very good/Good as one category and the remaining three as one category (Don't know will not be included). Question two on functional impairment will use all three answer categories (Don't know will not be included).

The outcome variables above (with 95% CIs) will be presented for the whole sample combined, and for the sample split on demographic and background variables 1-6 as outlined under the description of article I above. In addition, the outcome variables will be presented across the main outcome variables of article I: depression; anxiety; and PTSD (all binary). Furthermore, perceived general health will be reported across outcome variable one: pain in muscles and joints (3 categories) and general pain (3 categories); and outcome variable two: sleep difficulties (binary - insomnia vs. not). The number of participants contributing data to a specific statistics/analysis will be reported.

Article III:

Title: "Quality of life in adult Syrian refugees resettled in Norway between 2015 and 2017: a cross-sectional survey questionnaire study".

The main outcome variable of Article III will be quality of life (QoL) measured through The World Health Organization Quality of Life assessment (WHOQOL-BREF). All four domain-scores in the scale (physical health; psychological health; social relationships; and environment) will be used as outcome in analyses. In order to compare with relevant prior studies, the domain scores will be converted as needed according to the method described by the WHO. That is, results on quality of life will be presented in three different ways: as raw scores, converted to a 4-20 scale, and converted to a 0-100 scale. In order to be included in analysis for a certain domain, participants must have answered a minimum of six, five, two, and six items for the domains: physical health, psychological health, social relationships, and environment, respectively.

QoL scores (with standard deviation, SD, and 95% CIs) for the four domains will be presented for the whole sample combined, and for the sample split on demographic and background variables 1-6 as outlined under the description of article I above. In addition, QoL scores (with SD and 95% CIs) will be presented across the main outcome variables of article I: depression; anxiety; and PTSD (all binary); as well as the main outcome variables of article II: muscle/joint pain and general pain, both variables split into three categories: Not troubled (for all 5 items); Somewhat troubled (at least one item); Very troubled (at least one item); sleep difficulties (binary - insomnia vs. not); and perceived general health (binary for overall health, and three categories for functional impairment).

Furthermore QoL scores from REFUGE-I will be compared with scores from other refugee populations, and with QoL scores in the general population around the world. The number of participants contributing data to a specific statistics/analysis will be reported.

Ethical issues:

In the event that participation in the study triggers substantial adverse reactions in any of the participants, a help-line will be set up by the research team in collaboration with clinical personnel with experience on refugee mental health. Participants will be informed that they can send a text message to the help-line's phone number, and that the clinical personnel will call them back with an Arabic interpreter as soon as possible. Arrangements will be made with a professional Norwegian interpreter firm to ensure the availability of an interpreter within a reasonable time frame (hours). This service will be available during regular work hours. During off-hours and weekends, participants will be instructed to contact Norway's National out-of-hours medical service for immediate medical assistance and given the necessary information on how to do so.

ELIGIBILITY:
Inclusion Criteria:

* Syrian citizen who arrived to Norway as either resettlement refugee (quota refugee) or asylum seeker and asylum was granted/approved; or who arrived through the program: "Family immigration with a person who has protection (asylum) in Norway"
* Arrived to Norway between January 1, 2015 and December 31, 2017.
* Registered with a postal address in the Norwegian National Registry

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population comprises a random sample of 10 000 out of a total of 14350 resettled Syrians coming to Norway between January 1, 2015 and December 31, 2017 as: resettlement refugees (quota refugees), asylum seekers (approved asylum), or through family immigration (see Inclusion criteria). The sample was selected through simple random sampling (sampling fraction 0.7).
Sampling Method: Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2018-11-27 (Estimated); Primary Completion 2019-01-15 (Estimated); Study Completion 2019-01-15 (Estimated)

PRIMARY OUTCOMES:
Harvard Trauma Questionnaire (HTQ) | Collected as part of the survey questionnaire sent out to the sample of participants. Participants will have 6 weeks to answer and return the survey. Anticipated time frame for collection: November 27, 2018 to January 15, 2019.
  The first 16 items in the section on trauma symptoms (section IV) in the HTQ will be used to measure symptoms of posttraumatic stress disorder (PTSD) (Mollica et al., 1992; Shoeb, Weinstein, & Mollica, 2007). The selected 16 items are based on the criteria for PTSD diagnosis in the American Psychiatric Association's Diagnostic and Statistical Manual of mental disorders, version IV (DSM-IV). All 16 items have four categorical responses: Not at all; A little; Quite a bit; and Extremely; scored on a Likert-scale from 1 to 4, respectively. A mean item-score for the complete scale will be calculated (range: 1.0-4.0).
  As one of the main aims of REFUGE-I is to compare the prevalence of common mental health problems in resettled Syrian refugees in Norway to prevalences found in a parallel study in Sweden, REFUGE-I will use the same Arabic HTQ-version as was used in Sweden (Tinghög et al., 2017)
Hopkins Symptom Checklist (HSCL-25) | Collected as part of the survey questionnaire sent out to the sample of participants. Participants will have 6 weeks to answer and return the survey. Anticipated time frame for collection: November 27, 2018 to January 15, 2019.
  The HSCL-25 scale consists of 25 items and measures symptoms of anxiety and depression (Lavik, Hauff, Solberg, & Laake, 1999; Mollica, Wyshak, de Marneffe, Khuon, & Lavelle, 1987). Part I has 10 items for anxiety symptoms, and Part II has 15 items for depression symptoms. All items have four categorical responses: Not at all; A little; Quite a bit; and Extremely, scored on a Likert-scale from 1 to 4, respectively. Three mean scores are calculated: mean score for all 25 items; mean score for anxiety (average of the 10 anxiety items), and mean score for depression (average of the 15 depression items).
  As one of the main aims of REFUGE-I is to compare the prevalence of common mental health problems in resettled Syrian refugees in Norway to prevalences found in a parallel study in Sweden, REFUGE-I will use the same Arabic HSCL-version as was used in Sweden (Tinghög et al., 2017).
The World Health Organization Quality of Life assessment (WHOQOL-BREF) | Collected as part of the survey questionnaire sent out to the sample of participants. Participants will have 6 weeks to answer and return the survey. Anticipated time frame for collection: November 27, 2018 to January 15, 2019.
  WHOQOL-BREF is an abbreviated generic quality of life (QoL) scale developed through the World Health Organization (The WHOQOL Group, 1998). The scale contains 26 items. The first two items are stand-alone items aimed at measuring quality of life in general (item 1) and quality of life related to health (item 2). The other 24 items measure four different domains of quality of life: Physical health (7 items); Psychological health (6 items); Social relationships (3 items); and Environment (8 items). All items are scored on a 5-point Likert scale going from 1 (poor QoL) to 5 (high QoL). A tested and validated Arabic version of WHOQOL-BREF will be used (Ohaeri & Awadalla, 2009).

SECONDARY OUTCOMES:
Post-migration stress scale | Collected as part of the survey questionnaire sent out to the sample of participants. Participants will have 6 weeks to answer and return the survey. Anticipated time frame for collection: November 27, 2018 to January 15, 2019.
  Data on post-migration stress will be collected through the Post-migration stress scale developed by Malm et al (Malm, Tinghög, & Saboonchi, 2016). The complete scale consists of 24 items, all scored on a 5-point Likert scale ranging from 0 (Never) to 4 (Very often). Analyses will focus on seven questions thought to tap into the seven different domains of the Post-migration stress scale (for details, please see (Tinghög et al., 2017). The scale was translated into Arabic by the original research group (Malm et al., 2016)
Somatic pain: Likert scale | Collected as part of the survey questionnaire sent out to the sample of participants. Participants will have 6 weeks to answer and return the survey. Anticipated time frame for collection: November 27, 2018 to January 15, 2019.
  The questions on pain are based on The Tromsø Study, but slightly adapted to the study population of REFUGE-I (Andorsen, Ahmed, Emaus, & Klouman, 2016; "The Tromsø Study," n.d.). Participants will be asked about pain in muscles and joints in the last year, lasting for a minimum of 3 months, scored on a 3-point Likert scale (Not troubled; Somewhat troubled; and Very troubled) in the following 5 areas: Neck and shoulders; Arms or hands; Upper back, Lower back; and Hips, legs or feet. Similarly, using the same 3-point scale, participants will be asked about general pain in the following 5 areas: Stomach; Head; Genital area; Chest; and Other. The translation of the questions into Arabic was done by a professional translation bureau, then checked by two independent translators/interpreters. In addition, a thorough review was conducted by an Arabic speaking reference group from Syria.
Sleep difficulties | Collected as part of the survey questionnaire sent out to the sample of participants. Participants will have 6 weeks to answer and return the survey. Anticipated time frame for collection: November 27, 2018 to January 15, 2019.
  The Bergen Insomnia Scale will be used to investigate sleep difficulties (Pallesen et al., 2008). The six-item scale focuses on: problems falling asleep; extended awakenings during the night; early awakenings; feeling tired/fatigued/not rested after sleep; and overall dissatisfaction with sleep quality. All items are answered on a 8-point Likert scale going from 0 (No days in the week) to 7 (Every day during the week). A mean-item score will be calculated for the six questions combined (range: 0-7). The translation of the questions into Arabic was done by a professional translation bureau, then checked by two independent translators/interpreters. In addition, a thorough review was conducted by an Arabic speaking reference group from Syria.
Perceived general health | Collected as part of the survey questionnaire sent out to the sample of participants. Participants will have 6 weeks to answer and return the survey. Anticipated time frame for collection: November 27, 2018 to January 15, 2019.
  Two questions will used to measure perceived general health. Both questions are from the European Social Survey. Question one on overall health, "How is your health in general", has six answer categories: Very good; Good; Fair; Bad; Very bad; and Don't know. Question two, "Are you hampered in your daily activities in any way by any longstanding illness, or disability, infirmity or mental health problem?", taps into functional impairment and has four answer categories: No; Yes to some extent; Yes a lot; Don't know. The translation of the questions into Arabic was done by a professional translation bureau, then checked by two independent translators/interpreters. In addition, a thorough review was conducted by an Arabic speaking reference group from Syria.

OTHER OUTCOMES:
Refugee Trauma History Checklist (RTHC) | Collected as part of the survey questionnaire sent out to the sample of participants. Participants will have 6 weeks to answer and return the survey. Anticipated time frame for collection: November 27, 2018 to January 15, 2019.
  Data on potentially traumatic events experienced by study participants either before (premigration) or during (perimigration) their flight from their home will be collected using the Refugee Trauma History Checklist (RTHC) developed by Sigvardsdotter and colleagues (Sigvardsdotter et al., 2017). The checklist asks whether respondents have experienced eight potentially traumatic events either before or during their flight (separate scales for "before" vs "during"). In total, therefore, there are 16 items in the scale - 8 concerning premigration events and 8 concerning perimigration events, all answered on a binary outcome scale (Yes/No). The scale was translated into Arabic by the original research group (Sigvardsdotter et al., 2017).
Enhancing Recovery in Coronary Heart Disease (ENRICHD) Social Support Inventory (ESSI) | Collected as part of the survey questionnaire sent out to the sample of participants. Participants will have 6 weeks to answer and return the survey. Anticipated time frame for collection: November 27, 2018 to January 15, 2019.
  Data on social support will be collected using the first 6 items of the ENRICHD Social Support Inventory, ESSI (Mitchell et al., 2003). All 6 items are scored on a 5-point Likert scale going from 1 (None of the time) to 5 (All the time). The translation of the questions into Arabic was done by a professional translation bureau, then checked by two independent translators/interpreters. In addition, a thorough review was conducted by an Arabic speaking reference group from Syria.
Number of intrusive memories: | Collected as part of the survey questionnaire sent out to the sample of participants. Participants will have 6 weeks to answer and return the survey. Anticipated time frame for collection: November 27, 2018 to January 15, 2019.
  Intrusive memories (IMs) is described as: "relatively brief, vivid sensory impressions such as images, sounds, body sensations, tastes, or smells related to an event. They may or may not be triggered by something you are aware of, such as telling someone about what has happened to you or watching something on the news. Intrusive memories are not the same as deliberately thinking about a traumatic event or mulling it over". The definition is based on the DSM-V diagnostic manual and earlier research on Syrian refugees (Association & Others, 2013; Holmes et al., 2017). Participants will be asked if they experience IMs (Y/N), and if Yes, they will be asked how often they experience them (Less than monthly; Monthly; Weekly; Daily or almost daily; Several times each day; and how distressing they feel the IMs are on a scale from 0 to 10. The questions were translated following the same procedures as described under ESSI above.
Alcohol consumption | Collected as part of the survey questionnaire sent out to the sample of participants. Participants will have 6 weeks to answer and return the survey. Anticipated time frame for collection: November 27, 2018 to January 15, 2019.
  Participants will be asked the following four questions on alcohol (answer choices in parentheses):
  1. Whether they drink (Y/N).
  2. If yes, how often they drink (Never; Monthly or less; 2 to 4 times a month; 2 to 3 times a week; and 4 or more times a week).
  3. How many drinks containing alcohol they drink on a typical day when they drink (0; 1-2; 3-4; 5-6; 7-9; and 10 or more).
  4. How often they drink six or more drinks on one occasion (Never; Less than monthly; Monthly; Weekly; and Daily or almost daily).
  The translation of the questions into Arabic was done by a professional translation bureau, then checked by two independent translators/interpreters. In addition, a thorough review was conducted by an Arabic speaking reference group from Syria.

CONTACTS AND LOCATIONS:
Overall Officials: Arnfinn Andersen, Dr. Polit., Principal Investigator — Norwegian Center for Violence and Traumatic Stress Studies
Locations (1):
- Norwegian Center for Violence and Traumatic Stress Studies, Oslo, Norway

IPD SHARING:
Plan to Share IPD: Yes
The study's data sharing strategy has not yet been developed.
Time Frame: To be decided
Access Criteria: To be decided

REFERENCES:
- [Background] American Psychiatric Association. (2013). Diagnostic and statistical manual of mental disorders (5th ed.). Washington, DC: Author.
- [Background] Aziz IA, Hutchinson CV, Maltby J. Quality of life of Syrian refugees living in camps in the Kurdistan Region of Iraq. PeerJ. 2014 Nov 11;2:e670. doi: 10.7717/peerj.670. eCollection 2014. PMID 25401057
- [Background] BBC News. (2018, September 7). Why is there a war in Syria? BBC. Retrieved from https://www.bbc.com/news/world-middle-east-35806229
- [Background] Fazel M, Wheeler J, Danesh J. Prevalence of serious mental disorder in 7000 refugees resettled in western countries: a systematic review. Lancet. 2005 Apr 9-15;365(9467):1309-14. doi: 10.1016/S0140-6736(05)61027-6. PMID 15823380
- [Background] American Psychiatric Association. (1994). Diagnostic and statistical manual of mental disorders (4th ed.). Washington, DC: Author.
- [Background] Holmes EA, Ghaderi A, Eriksson E, Lauri KO, Kukacka OM, Mamish M, James EL, Visser RM. 'I Can't Concentrate': A Feasibility Study with Young Refugees in Sweden on Developing Science-Driven Interventions for Intrusive Memories Related to Trauma. Behav Cogn Psychother. 2017 Mar;45(2):97-109. doi: 10.1017/S135246581600062X. PMID 28229806
- [Background] Lavik, N. J., Hauff, E., Solberg, Ø., & Laake, P. (1999). The use of self-reports in psychiatric studies of traumatized refugees: Validation and analysis of HSCL-25. Nordic Journal of Psychiatry, 53(1), 17-20. https://doi.org/10.1080/080394899426666
- [Background] Malm, A., Tinghög, P., & Saboonchi, F. (2016). Post-migration stress among refugees - development of a new scale and associations with wellbeing. European Health Psychologist, 18(S), 651. Retrieved from http://www.ehps.net/ehp/index.php/contents/article/view/2004
- [Background] Mitchell PH, Powell L, Blumenthal J, Norten J, Ironson G, Pitula CR, Froelicher ES, Czajkowski S, Youngblood M, Huber M, Berkman LF. A short social support measure for patients recovering from myocardial infarction: the ENRICHD Social Support Inventory. J Cardiopulm Rehabil. 2003 Nov-Dec;23(6):398-403. doi: 10.1097/00008483-200311000-00001. No abstract available. PMID 14646785
- [Background] Mollica RF, Caspi-Yavin Y, Bollini P, Truong T, Tor S, Lavelle J. The Harvard Trauma Questionnaire. Validating a cross-cultural instrument for measuring torture, trauma, and posttraumatic stress disorder in Indochinese refugees. J Nerv Ment Dis. 1992 Feb;180(2):111-6. PMID 1737972
- [Background] Mollica RF, Wyshak G, de Marneffe D, Khuon F, Lavelle J. Indochinese versions of the Hopkins Symptom Checklist-25: a screening instrument for the psychiatric care of refugees. Am J Psychiatry. 1987 Apr;144(4):497-500. doi: 10.1176/ajp.144.4.497. PMID 3565621
- [Background] Morina N, Akhtar A, Barth J, Schnyder U. Psychiatric Disorders in Refugees and Internally Displaced Persons After Forced Displacement: A Systematic Review. Front Psychiatry. 2018 Sep 21;9:433. doi: 10.3389/fpsyt.2018.00433. eCollection 2018. PMID 30298022
- [Background] Shoeb M, Weinstein H, Mollica R. The Harvard trauma questionnaire: adapting a cross-cultural instrument for measuring torture, trauma and posttraumatic stress disorder in Iraqi refugees. Int J Soc Psychiatry. 2007 Sep;53(5):447-63. doi: 10.1177/0020764007078362. PMID 18018666
- [Background] Sigvardsdotter E, Nilsson H, Malm A, Tinghog P, Gottvall M, Vaez M, Saboonchi F. Development and Preliminary Validation of Refugee Trauma History Checklist (RTHC)-A Brief Checklist for Survey Studies. Int J Environ Res Public Health. 2017 Oct 4;14(10):1175. doi: 10.3390/ijerph14101175. PMID 28976937
- [Background] Statistics Norway (SSB). (n.d.). Retrieved October 5, 2018, from https://www.ssb.no/en
- [Background] Development of the World Health Organization WHOQOL-BREF quality of life assessment. The WHOQOL Group. Psychol Med. 1998 May;28(3):551-8. doi: 10.1017/s0033291798006667. PMID 9626712
- [Background] Tinghog P, Malm A, Arwidson C, Sigvardsdotter E, Lundin A, Saboonchi F. Prevalence of mental ill health, traumas and postmigration stress among refugees from Syria resettled in Sweden after 2011: a population-based survey. BMJ Open. 2017 Dec 29;7(12):e018899. doi: 10.1136/bmjopen-2017-018899. PMID 29289940
- [Background] United Nations High Commissioner for Refugees. (2018). Syria emergency. Retrieved October 5, 2018, from http://www.unhcr.org/syria-emergency.html
- [Background] World Health Organization. Division of Mental Health. (1996). WHOQOL-BREF : introduction, administration, scoring and generic version of the assessment : field trial version, December 1996. Geneva : World Health Organization. http://www.who.int/iris/handle/10665/63529
- [Derived] Nissen A, Hynek KA, Scales D, Hilden PK, Straiton M. Chronic pain, mental health and functional impairment in adult refugees from Syria resettled in Norway: a cross-sectional study. BMC Psychiatry. 2022 Aug 24;22(1):571. doi: 10.1186/s12888-022-04200-x. PMID 36002823
- [Derived] Nissen A, Cauley P, Saboonchi F, Andersen A, Solberg O. Cohort profile: Resettlement in Uprooted Groups Explored (REFUGE)-a longitudinal study of mental health and integration in adult refugees from Syria resettled in Norway between 2015 and 2017. BMJ Open. 2020 Jul 1;10(7):e036101. doi: 10.1136/bmjopen-2019-036101. PMID 32611742